CLINICAL TRIAL: NCT06561581
Title: Acuity Functional Impact and Implementation Outcomes Evaluation
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Experiad LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Acuity-Study-1
Record Dates: First submitted 2024-08-09; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acuity-Basic (Other)
  Interventions: Behavioral: Acuity
- Acuity-Enhanced (Experimental)
  Interventions: Behavioral: Acuity

INTERVENTIONS:
Behavioral: Acuity — Enhancement to Motivity product for clinical decision support
  Other Names: Motivity

SUMMARY:
This study will test feature enhancements to a behavioral therapy data collection software (Motivity) that will add a new clinical decision support module, called Acuity. Acuity is a Quality Improvement (QI) intervention targeted at Behavior Analysts (BAs) and Behavior Technicians (BTs) that aims to improve the delivery of autism behavioral therapy. Subjects will be staff recruited from existing Motivity customers.

DETAILED DESCRIPTION:
Acuity is intended to provide significant improvements in treatment planning, progress tracking, trend monitoring, and dosage management. If successful, Acuity will provide Applied Behavior Analysis (ABA) practitioners with a higher level of real-time insight into their clinical data, enabling more efficient and productive treatment. Research has shown that first-generation systems fall short in supporting overworked BAs who are overwhelmed with data. Acuity will address critical shortfalls by enabling more agile corrective actions and data-driven planning across multiple aspects of treatment, providing practitioners with new levels of rigorous, real-time insight into their clinical data. Acuity will help BAs establish and adhere to realistic treatment timelines, and will proactively alert the BA to noteworthy trends in the data as they occur, such as learner performance issues, missed dosages, and significant changes in tracked behaviors. In doing so, Acuity will support more responsive and effective treatment.

ELIGIBILITY:
Inclusion Criteria:

* Behavior Analysts and Behavior Technicians treating kids with autism
* Must be employed by one of the autism treatment clinics that have agreed to participate in the study.
* Must be employed by Experiad customers who are using Motivity software as part of their practice.

Exclusion Criteria:

* All people not listed above

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with improved estimation of Trials to Criterion and Time (days) to Criterion | through study completion, expected to be 18 months from the start of retroactive observation period
  Does Acuity make initial timeline estimates for sets of targets more accurate?
Increased frequency of changes to programs and prescribed dosages, resulting in reduced Trials to Criterion and Time to Criterion. | through study completion, expected to be 18 months from the start of retroactive observation period
  Does Acuity result in corrective action being taken more quickly for programs that are off schedule or targets that are exhibiting performance issues?
Increased adherence to prescribed dosage | through study completion, expected to be 18 months from the start of retroactive observation period
  Does Acuity result in increased adherence to prescribed dosage, as measured by system
Number of participants who find Acuity and its components practical and possible to use, assessed by qualitative measures and system usage tracking | at the end of the study, expected to be 18 months from the start of retroactive observation period
  Feasibility - To what extent are Acuity and its components practical or possible to use?
Proportion of clinics and providers that actively use Acuity, assessed by system usage tracking. | at the end of the study, expected to be 18 months from the start of retroactive observation period
  Adoption - What proportion of clinics and providers are willing to use Acuity and how well do they represent the population of clinics and providers?
Number of BAs & BTs who utilize Acuity as intended to provide learners with accurate treatment plans, and achieve expected results, as measured by system usage and qualitative assessment. | at the end of the study, expected to be 18 months from the start of retroactive observation period
  Fidelity - the degree to which BAs and BTs use the system as expected, including dosage adherence, treatment planning accuracy, and timely protocol modification.
Majority of BAs and BTs rate Acuity and its components as attractive, agreeable, or palatable. | at the end of the study, expected to be 18 months from the start of retroactive observation period
  Acceptability, as measured by SUS score and SUS Items 1, 5, 6 & 8 collected via online survey at the end of O0 & O1 from both arms.
Frequency at which Acuity and its components are rated as suitable, fitting, or proper for achieving the goals set forth in treatment plans, as measured by surveys. | at the end of the study, expected to be 18 months from the start of retroactive observation period
  Appropriateness - Same measures captured for all primary & secondary research questions in the Functional Impact Evaluation. Brief online survey with Likert scaled items focused on the providers' assessment of how well Acuity and its components are matched to the challenges of planning and executing Treatment Plans.

CONTACTS AND LOCATIONS:
Locations (1):
- Experiad LLC, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No